CLINICAL TRIAL: NCT01457430
Title: Open Label, Multicenter Study to Evaluate Efficacy, Safety and Tolerability of a Self-Administered Subcutaneous Formulation of Icatibant for the Treatment of Acute Attacks of Hereditary Angioedema (IHA)
Brief Title: Efficacy, Safety and Tolerability of Icatibant for the Treatment of HAE
Acronym: IHA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shire Human Genetic Therapies, Inc. (Industry)
Responsible Party: Principal Investigator, Aleena Banerji, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011P001768
Record Dates: First submitted 2011-10-13; First posted 2011-10-24 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — icatibant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icatibant (Experimental): Open-label study
  Interventions: Drug: Icatibant

INTERVENTIONS:
Drug: Icatibant — 30 mg subcutaneous dose of Icatibant
  Other Names: Firazyr

SUMMARY:
The investigators propose a study to evaluate the safety, local tolerability, convenience, and efficacy of self-administered Icatibant for the treatment of acute attacks of hereditary angioedema. The investigators believe that self administration with Icatibant for treatment of an acute attack of angioedema will not change the time to complete or near complete resolution of symptoms compared to treatment with Icatibant in a medical facility.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 18 years of age at the time of informed consent
2. Documented diagnosis of hereditary angioedema Type I or II based on ALL of the following criteria:

   * Family and/or medical history
   * Characteristic attack manifestations, recurrent attacks
   * Historical low C4, normal C1q and either low C1-INH or low C1INH function
3. Women of childbearing potential must use consistently and correctly a highly effective, adequate method of birth control (failure rate less than 1% per year), sexual abstinence or have a vasectomised partner during the duration of the study. Hormonal contraception can be continued if verified by a physician that it doesn't affect the course of hereditary angioedema attacks.
4. Mental and physical condition allowing patients to complete baseline assessment, to self-administer Icatibant and to follow other study procedures.
5. Ability to provide signed written informed consent after all aspects of the study have been explained and discussed with the patient.

Exclusion Criteria:

1. Participation in a clinical therapeutic trial of another investigational medicinal product within the past month (except a previous Icatibant study).
2. Diagnosis of angioedema other than Type I or Type II hereditary angioedema.
3. Evidence of symptomatic coronary artery disease based on medical history, in particular, unstable angina pectoris or severe coronary heart disease.
4. Congestive heart failure (NYHA Class 3 and 4).
5. Stroke within the past 6 months.
6. Treatment with angiotensin converting enzyme inhibitor.
7. Pregnancy and/or breast-feeding.
8. In the opinion of the investigator: mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study.
9. In the opinion of the investigator: unlikely to comply with the protocol, for example, uncooperative attitude, inability to return for follow-up visits, or unlikely to complete the study for any reason.
10. In the opinion of the investigator: inability to complete the patient diary, manage study medication or self-administration of an injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleena Banerji, M.D., Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - San Diego Veterans Affairs Medical Center, La Jolla, California
  - UCLA - David Geffen School of Medicine, Los Angeles, California
  - Institute for Allergy and Asthma, Wheaton, Maryland
  - Penn State University, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided
The data is under review for publication but individual data will likely not be available

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Icatibant
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Icatibant
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 41 [19 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete or Near Complete Resolution From Onset of Symptoms
Description: Time of onset of HAE attack, time icatibant was administered, and time to complete relief of symptoms were recorded in minutes. Time to complete relief of symptoms was defined as time from onset of symptoms to complete or near complete resolution as reported by the patient.
Time Frame: Time to complete or near complete resolution of symptoms as reported by the patient, an expected average of 8-10 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Icatibant Treatment With Health Care Provider: Icatibant: 30 mg subcutaneous dose of Icatibant given to treat an acute attack of HAE by a health care provider.
- Icatibant Treatment by Self Administration: Icatibant: 30 mg subcutaneous dose of Icatibant given to treat an acute attack of HAE by self administration.
Arm/Group | Icatibant Treatment With Health Care Provider | Icatibant Treatment by Self Administration
Number analyzed (Participants) | 19 | 19
minutes | 735 [339 to 1563] | 377 [220 to 618]

2. Secondary Outcome: Percent Change in VAS Scores
Description: Baseline, 4 hours VAS scale ranges from 0-100 with 0 being the lowest severity and 100 being the highest severity
Time Frame: Percent Change in VAS Score from Baseline to 4 Hours
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Icatibant Treatment With Health Care Provider | Icatibant Treatment by Self Administration
Number analyzed (Participants) | 19 | 19
percent change | -97 [-100 to -73] | -96 [-100 to -80]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the study.
Description: Adverse events were assessed out of total attacks, not total participants. There were 78 HAE attacks with data collected and recorded on adverse events.
Arm/Group | Icatibant
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 4/78
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icatibant (N=78)
Fatigue (Blood and lymphatic system disorders) | 1 (1)
Fever (Blood and lymphatic system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
All adverse events were recorded and assessed out of total attacks, not total participants. There were 78 HAE attacks; 4 adverse events were identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No